CLINICAL TRIAL: NCT03663699
Title: Increasing Physical Activity Among Adolescents With Motivational High-Intensity Training Through a Cutting-Edge Gaming Platform
Brief Title: Gaming and Training Combined to Help Adolescents Get More Physically Active
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: grunnet COVID-19 pandemien då vi haft hög drop-out og vanskelig att rekruttere
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/633
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Sedentary Lifestyle
Keywords: Exercise Therapy; Physical Fitness; Games, Recreational; Children; Adolescents; Healthy Lifestyle; Exercise Test
MeSH Terms: conditions — Sedentary Behavior | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming (Experimental): 24 week access to the exergaming platform PlayPulse
  Interventions: Behavioral: Exergaming
- Control (No Intervention): Asked to continue with their normal daily routine

INTERVENTIONS:
Behavioral: Exergaming — free access to the exergaming platform PlayPulse for 24 weeks
  Other Names: PlayPulse
  Arms: Exergaming

SUMMARY:
The purpose of this study is to investigate if playing a newly developed videogame that requires physical activity (e.g. exergame), leads to increased physical activity and health benefits in children and adolescents who do not regularly participate in endurance training. Health benefits will be expressed in physical fitness (maximal oxygen consumption), blood markers of a healthy heart, body composition and objectively measured physical activity. Gaming frequency of the participants will be registered throughout the 24 week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Not regularly participating in endurance training
* Sedentary (<60 mins daily moderate/vigorous intensity physical activity)
* Play video games > 10 hours/week (self-reported)
* Able to ride a bike for up to 60 minutes

Exclusion Criteria:

* Known cardiovascular disease
* Type I diabetes

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
VO2max | 12 weeks
  Maximal Aerobic Capacity
VO2max | 24 weeks
  Maximal Aerobic Capacity

SECONDARY OUTCOMES:
Change in daily average energy expenditure | Baseline, 12 and 24 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 12 weeks and 24 weeks.
Change in daily time in sedentary activity (<3.0 metabolic equivalents =METs) | Baseline, 12 and 24 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 12 weeks and 24 weeks.
Change in daily time in moderate intensity activity (3.0-6.0 metabolic equivalents = METs) | Baseline, 12 and 24 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 12 weeks and 24 weeks.
Change in daily time in vigorous intensity activity (6.0-9.0 metabolic equivalents = METs) | Baseline, 12 and 24 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 12 weeks and 24 weeks.
Change in daily time in very vigorous intensity activity (>9.0 metabolic equivalents = METs) | Baseline, 12 and 24 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 12 weeks and 24 weeks.
Change in daily average total physical activity duration | Baseline, 12 and 24 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 12 weeks and 24 weeks.
Change in daily average number of steps | Baseline, 12 and 24 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period, 12 weeks and 24 weeks.
Bioelectrical impedance | 12 and 24 weeks
  Body composition assessed using bioelectrical impedance analysis (InBody 720)
systolic Blood Pressure | 12 and 24 weeks
Diastolic Blood Pressure | 12 and 24 weeks
Fasting circulating glucose, as blood marker of cardiometabolic health | 24 weeks
Lipid profile, as blood marker of cardiometabolic health | 24 weeks
Circulating insulin concentration, as blood marker of cardiometabolic health | 24 weeks
HbA1c from blood samples | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No